CLINICAL TRIAL: NCT00452400
Title: Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study to Assess the Efficacy and Safety of 4 Weeks of Treatment of Orally Inhaled BI 1744 CL (3 - 4 Doses) Delivered by the Respimat® Inhaler in Patients With COPD
Brief Title: Efficacy and Safety of 4 Weeks Treatment With Inhaled BI 1744 CL in Patients With COPD.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1222.5
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

INTERVENTIONS:
Drug: BI 1744CL

SUMMARY:
The primary objective of this study is to determine the optimum dose(s) of BI 1744 CL inhalation solution delivered by the Respimat® inhaler for four weeks in patients with chronic obstructive pulmonary disease (COPD). The selection of the optimum dose(s) will be based on bronchodilator efficacy (how well it helps your breathing), safety evaluations and pharmacokinetic evaluations (the amount of the medication found in your blood).

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent consistent with ICH-GCP guidelines prior to participation in the trial, which includes medication washout and restrictions
2. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

   Patients must have relatively stable, moderate to severe airway obstruction with a post-bronchodilator FEV1  30% of predicted normal and < 80% of predicted normal and a post-bronchodilator FEV1 / FVC < 70% at Visit 1
3. Male or female patients, 40 years of age or older
4. Patients must be current or ex-smokers with a smoking history of more than 10 pack years. Patients who have never smoked cigarettes must be excluded
5. Patients must be able to perform technically acceptable pulmonary function tests and PEFR measurements, and must be able to maintain records (Patient Daily e-Diary) during the study period as required in the protocol
6. Patients must be able to inhale medication in a competent manner from the Respimat® inhaler and from a metered dose inhaler (MDI).

Exclusion Criteria:

Selection of relevant exclusion criteria:

1. Patients with a history of asthma or a total blood eosinophil count 600/mm3.
2. Patients with any of the following conditions:

   * a diagnosis of thyrotoxicosis
   * a diagnosis of paroxysmal tachycardia (>100 beats per minute)
   * a marked baseline prolongation of QT/QTc interval (e.g. repeated demonstration of a QTc interval > 450 ms).
   * a history of additional risk factors for Torsade de Pointes (TdP) (e.g. heart failure, hypokalemia, family history of Long QT Syndrome)
3. Patients with any of the following conditions:

   * a history of myocardial infarction within 1 year of screening visit (Visit 1)
   * a diagnosis of clinically relevant cardiac arrhythmia
   * known active tuberculosis
   * a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years (patients with treated basal cell carcinoma are allowed)
   * a history of life-threatening pulmonary obstruction
   * a history of cystic fibrosis
   * clinically evident bronchiectasis
   * a history of significant alcohol or drug abuse
4. Patients who have undergone thoracotomy with pulmonary resection
5. Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy during clinic visits
6. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the Screening Visit (Visit 1) or patients who are currently in a pulmonary rehabilitation program
7. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to Screening Visit (Visit 1)
8. Pregnant or nursing women
9. Women of childbearing potential not using a highly effective method of birth control
10. Patients who have previously been randomized in this study or are currently participating in another study
11. Patients who are unable to comply with medication restrictions.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (42):
- United States (22):
  - 1222.5.03 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1222.5.07 Boehringer Ingelheim Investigational Site, Lakewood, California
  - 1222.5.14 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1222.5.13 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1222.5.17 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1222.5.18 Boehringer Ingelheim Investigational Site, Stamford, Connecticut
  - 1222.5.15 Boehringer Ingelheim Investigational Site, Panama City, Florida
  - 1222.5.04 Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - 1222.5.22 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 1222.5.11 Boehringer Ingelheim Investigational Site, Reno, Nevada
  - 1222.5.24 Boehringer Ingelheim Investigational Site, New York, New York
  - 1222.5.12 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 1222.5.10 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 1222.5.05 Boehringer Ingelheim Investigational Site, Hershey, Pennsylvania
  - 1222.5.02 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1222.5.08 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1222.5.19 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1222.5.06 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1222.5.21 Boehringer Ingelheim Investigational Site, Kileen, Texas
  - 1222.5.01 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1222.5.23 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1222.5.20 Boehringer Ingelheim Investigational Site, Tacoma, Washington
- Canada (10):
  - 1222.5.039 St. Boniface General Hospital & Health Science Centre, Winnipeg, Manitoba
  - 1222.5.032 Division of Respirology, Halifax, Nova Scotia
  - 1222.5.038 Courtice Health Centre, Courtice, Ontario
  - 1222.5.037 Kingston General Hospital, Kingston, Ontario
  - 1222.5.031 Alpha Medical Research Inc., Mississauga, Ontario
  - 1222.5.034 Pulmonary Care Clinic and Research Centre, Toronto, Ontario
  - 1222.5.040 Respiratory Research Lab, Toronto, Ontario
  - 1222.5.033 Centre de Recherche Clinique -CHUS, Sherbrooke, Quebec
  - 1222.5.035 Hopital Laval, Ste-Foy, Quebec
  - 1222.5.036 Department of Respiratory Medicine, Saskatoon, Saskatchewan
- Germany (6):
  - 1222.5.046 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.5.049 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.5.052 Boehringer Ingelheim Investigational Site, Gauting
  - 1222.5.051 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1222.5.047 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 1222.5.048 Boehringer Ingelheim Investigational Site, Wiesbaden
- Netherlands (4):
  - 1222.5.058 Boehringer Ingelheim Investigational Site, Almelo
  - 1222.5.056 Boehringer Ingelheim Investigational Site, Breda
  - 1222.5.059 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1222.5.057 Boehringer Ingelheim Investigational Site, Heerlen

REFERENCES:
- [Derived] Maleki-Yazdi MR, Beck E, Hamilton AL, Korducki L, Koker P, Fogarty C. A randomised, placebo-controlled, Phase II, dose-ranging trial of once-daily treatment with olodaterol, a novel long-acting beta2-agonist, for 4 weeks in patients with chronic obstructive pulmonary disease. Respir Med. 2015 May;109(5):596-605. doi: 10.1016/j.rmed.2015.02.012. Epub 2015 Mar 3. PMID 25829298

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 409 patients were enrolled to the study, however 4 patients were assigned incorrect medication, so these patients were re-randomised, so only 405 patients actually started the study.
Groups:
- Placebo: Matching Placebo delivered by the Respimat Inhaler.
- Olo 2 mcg qd: Olodaterol 2 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 5 mcg qd; Olo 10 mcg qd: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 20 mcg qd: Olodaterol 20 mcg qd (morning) delivered by the Respimat Inhaler.
Period: Overall Study
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Started | 79 | 81 | 80 | 86 | 79
Completed | 74 | 80 | 73 | 85 | 76
Not Completed | 5 | 1 | 7 | 1 | 3
Not completed — Adverse Event | 1 | 1 | 5 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0
Not completed — Other reasons not listed above | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated set includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd | Total
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79 | 405
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.66 (9.74) | 63.81 (8.63) | 63.25 (9.47) | 63.55 (7.92) | 63.19 (9.00) | 63.30 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 39 | 24 | 35 | 33 | 171
  Male | 39 | 42 | 56 | 51 | 46 | 234

OUTCOME MEASURES:

1. Primary Outcome: Trough FEV1 Response After 4 Weeks
Description: Trough FEV1 is defined as the mean of the two FEV1 values (performed at -1 hour and -10 minutes prior to test-drug inhalation) at the end of the dosing interval, 24 hours post-drug administration. Trough FEV1 response is defined as the change from baseline in trough FEV1. Baseline FEV1 is the mean of the two pre-treatment FEV1 values measured at Visit 2 (- 1 hour and - 10 minutes) prior to administration of the first dose of study medication.
Time Frame: Baseline and 4 weeks
Population: Full analysis set (FAS) is defined as all randomized patients who received at least one dose of treatment and had baseline data for at least one endpoint.
Measure: Least Squares Mean (Standard Error); unit: Liter
Groups:
- Olo 5 mcg qd: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | -0.014 (0.021) | 0.046 (0.021) | 0.082 (0.021) | 0.109 (0.021) | 0.118 (0.021)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0233, ANCOVA; Based on an analysis of covariance with terms for baseline, treatment and center (center random, all other effects fixed); Mean Difference (Final Values) = 0.061, 95% CI [0.008 to 0.113], Standard Error of Mean 0.027 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0003, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.097, 95% CI [0.044 to 0.149], Standard Error of Mean 0.027 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.123, 95% CI [0.072 to 0.175], Standard Error of Mean 0.026 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.132, 95% CI [0.080 to 0.185], Standard Error of Mean 0.027 — Olo 20 mcg qd minus Placebo

2. Secondary Outcome: Trough FEV1 Response After 1 Week
Description: as for outcome 1
Time Frame: Baseline and 1 week
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | -0.029 (0.019) | 0.059 (0.018) | 0.108 (0.019) | 0.099 (0.018) | 0.140 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0004, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.088, 95% CI [0.039 to 0.137], Standard Error of Mean 0.025 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.137, 95% CI [0.088 to 0.186], Standard Error of Mean 0.025 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.128, 95% CI [0.080 to 0.176], Standard Error of Mean 0.024 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.169, 95% CI [0.120 to 0.218], Standard Error of Mean 0.025 — Olo 20 mcg qd minus Placebo

3. Secondary Outcome: Trough FEV1 Response After 2 Weeks
Description: as for outcome 1
Time Frame: Baseline and 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | -0.023 (0.020) | 0.062 (0.020) | 0.099 (0.020) | 0.102 (0.020) | 0.105 (0.020)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0011, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.085, 95% CI [0.034 to 0.136], Standard Error of Mean 0.026 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.121, 95% CI [0.070 to 0.173], Standard Error of Mean 0.026 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.125, 95% CI [0.075 to 0.175], Standard Error of Mean 0.026 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.128, 95% CI [0.077 to 0.179], Standard Error of Mean 0.026 — Olo 20 mcg qd minus Placebo

4. Secondary Outcome: Trough FVC Response After 1 Week
Description: Trough FVC was defined as the mean of the two values obtained at 1 hour and 10 minutes prior to the pulmonary function test maneuver. Response is defined as change from the baseline value. Study baseline FVC was defined as the mean of the available pre-dose FVC values prior to the first dose of randomized treatment.
Time Frame: Baseline and 1 week
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | -0.020 (0.033) | 0.090 (0.033) | 0.154 (0.033) | 0.149 (0.032) | 0.151 (0.033)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0127, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.110, 95% CI [0.024 to 0.197], Standard Error of Mean 0.044 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.174, 95% CI [0.087 to 0.261], Standard Error of Mean 0.044 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.170, 95% CI [0.084 to 0.255], Standard Error of Mean 0.043 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.171, 95% CI [0.084 to 0.258], Standard Error of Mean 0.044 — Olo 20 mcg qd minus Placebo

5. Secondary Outcome: Trough FVC Response After 2 Weeks
Description: as for outcome 4
Time Frame: Baseline and 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | -0.000 (0.040) | 0.090 (0.040) | 0.171 (0.040) | 0.149 (0.039) | 0.148 (0.040)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0836, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.090, 95% CI [-0.012 to 0.192], Standard Error of Mean 0.052 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0011, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.171, 95% CI [0.068 to 0.274], Standard Error of Mean 0.052 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0037, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.150, 95% CI [0.049 to 0.250], Standard Error of Mean 0.051 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0047, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.148, 95% CI [0.046 to 0.251], Standard Error of Mean 0.052 — Olo 20 mcg qd minus Placebo

6. Secondary Outcome: Trough FVC Response After 4 Weeks
Description: as for outcome 4
Time Frame: Baseline and 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | -0.026 (0.040) | 0.068 (0.040) | 0.136 (0.040) | 0.146 (0.039) | 0.153 (0.040)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0695, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.094, 95% CI [-0.008 to 0.195], Standard Error of Mean 0.051 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0018, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.162, 95% CI [0.061 to 0.264], Standard Error of Mean 0.052 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0008, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.172, 95% CI [0.072 to 0.272], Standard Error of Mean 0.051 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0006, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.179, 95% CI [0.077 to 0.281], Standard Error of Mean 0.052 — Olo 20 mcg qd minus Placebo

7. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-6 h (AUC 0-6h) Response at Week 4
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of randomized treatment. Means are adjusted using a model with treatment (trt), baseline as fixed effects and centre as random effect. FEV1 AUC 0-6h was calculated from 0-6 hours post-dose using the trapezoidal rule, divided by the observation time (6h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on first day of randomized treatment (baseline) and 30 min, 1h, 2h, 3h, 4h, 5h, 6h relative to dose at Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | 0.013 (0.025) | 0.154 (0.024) | 0.175 (0.025) | 0.226 (0.024) | 0.228 (0.025)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.141, 95% CI [0.078 to 0.204], Standard Error of Mean 0.032 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.162, 95% CI [0.099 to 0.225], Standard Error of Mean 0.032 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.213, 95% CI [0.151 to 0.275], Standard Error of Mean 0.031 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.214, 95% CI [0.151 to 0.277], Standard Error of Mean 0.032 — Olo 20 mcg qd minus Placebo

8. Secondary Outcome: Peak FEV1 (0-3h) Response After 4 Weeks
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of randomized treatment. Peak FEV1 (0-3h) values were obtained within 0 - 3 hours after treatment. Means are adjusted using a mixed effects model with baseline, treatment and centre (centre random, all other effects fixed).
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to 30 min, 1 h, 2 h, and 3 h relative to dose after 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | 0.078 (0.026) | 0.242 (0.026) | 0.247 (0.026) | 0.295 (0.025) | 0.303 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.164, 95% CI [0.097 to 0.231], Standard Error of Mean 0.034 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.169, 95% CI [0.102 to 0.237], Standard Error of Mean 0.034 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.218, 95% CI [0.152 to 0.284], Standard Error of Mean 0.034 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.225, 95% CI [0.157 to 0.292], Standard Error of Mean 0.034 — Olo 20 mcg qd minus Placebo

9. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-6 h (AUC 0-6h) Response at Week 4
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values prior to the first dose of randomized treatment. Means are adjusted using a model with treatment (trt), baseline as fixed effects and centre as random effect. FVC AUC 0-6h was calculated from 0-6 hours post-dose using the trapezoidal rule, divided by the observation time (6h) to report in litres.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | 0.009 (0.044) | 0.271 (0.043) | 0.292 (0.044) | 0.320 (0.042) | 0.313 (0.044)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.262, 95% CI [0.150 to 0.373], Standard Error of Mean 0.057 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.283, 95% CI [0.171 to 0.395], Standard Error of Mean 0.057 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.311, 95% CI [0.201 to 0.421], Standard Error of Mean 0.056 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.304, 95% CI [0.192 to 0.416], Standard Error of Mean 0.057 — Olo 20 mcg qd minus Placebo

10. Secondary Outcome: Peak FVC (0-3h) Response After 4 Weeks
Description: Peak (0-3h) will be the maximum post-dose value during the first 3 hours. Response is defined as change from the baseline value. Study baseline FVC was defined as the mean of the available pre-dose FVC values prior to the first dose of randomized treatment.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | 0.152 (0.046) | 0.440 (0.046) | 0.432 (0.046) | 0.449 (0.044) | 0.438 (0.046)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.288, 95% CI [0.167 to 0.409], Standard Error of Mean 0.061 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.280, 95% CI [0.159 to 0.401], Standard Error of Mean 0.062 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.297, 95% CI [0.178 to 0.416], Standard Error of Mean 0.061 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.286, 95% CI [0.164 to 0.407], Standard Error of Mean 0.062 — Olo 20 mcg qd minus Placebo

11. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-3 h (AUC 0-3h) Response at Day 1
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of randomized treatment. Means are adjusted using a model with treatment (trt), baseline as fixed effects and centre as random effect. FEV1 AUC 0-3h was calculated from 0-3 hours postdose using the trapezoidal rule, divided by the observation time (3h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on first day of randomized treatment (baseline) and 30 min, 1h, 2h, 3h relative to dose at day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | 0.031 (0.017) | 0.165 (0.017) | 0.203 (0.017) | 0.236 (0.017) | 0.234 (0.017)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.133, 95% CI [0.090 to 0.176], Standard Error of Mean 0.022 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.172, 95% CI [0.128 to 0.215], Standard Error of Mean 0.022 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 0.204, 95% CI [0.162 to 0.247], Standard Error of Mean 0.022 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 0.203, 95% CI [0.159 to 0.246], Standard Error of Mean 0.022 — Olo 20 mcg qd minus Placebo

12. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-3 h (AUC 0-3h) Response at Week 1
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of randomized treatment. Means are adjusted using a model with treatment (trt), baseline as fixed effects and centre as random effect. FEV1 AUC 0-3h was calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time (3h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on first day of randomized treatment (baseline) and 30 min, 1h, 2h, 3h relative to dose at Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | -0.000 (0.022) | 0.186 (0.022) | 0.215 (0.022) | 0.218 (0.021) | 0.247 (0.022)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.187, 95% CI [0.131 to 0.243], Standard Error of Mean 0.028 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.215, 95% CI [0.159 to 0.271], Standard Error of Mean 0.029 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.218, 95% CI [0.163 to 0.273], Standard Error of Mean 0.028 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.247, 95% CI [0.191 to 0.304], Standard Error of Mean 0.029 — Olo 20 mcg qd minus Placebo

13. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-3 h (AUC 0-3h) Response at Week 2
Description: as for outcome 12
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on first day of randomized treatment (baseline) and 30 min, 1h, 2h, 3h relative to dose at Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | 0.006 (0.024) | 0.166 (0.024) | 0.200 (0.024) | 0.209 (0.023) | 0.211 (0.024)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.159, 95% CI [0.100 to 0.219], Standard Error of Mean 0.030 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.194, 95% CI [0.134 to 0.253], Standard Error of Mean 0.030 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.203, 95% CI [0.144 to 0.262], Standard Error of Mean 0.030 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.204, 95% CI [0.145 to 0.264], Standard Error of Mean 0.030 — Olo 20 mcg qd minus Placebo

14. Secondary Outcome: Peak FEV1 (0-3h) Response At Day 1
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of randomized treatment. Peak FEV1 (0-3h) values were obtained within 0 - 3 hours after treatment.Means are adjusted using a mixed effects model with baseline,treatment and centre (centre random, all other effects fixed).
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to 30 min, 1 h, 2 h, and 3 h relative to dose at day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | 0.104 (0.021) | 0.259 (0.021) | 0.288 (0.021) | 0.335 (0.020) | 0.335 (0.021)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.155, 95% CI [0.101 to 0.209], Standard Error of Mean 0.027 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.185, 95% CI [0.131 to 0.239], Standard Error of Mean 0.027 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.231, 95% CI [0.178 to 0.284], Standard Error of Mean 0.027 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.231, 95% CI [0.177 to 0.286], Standard Error of Mean 0.028 — Olo 20 mcg qd minus Placebo

15. Secondary Outcome: Peak FEV1 (0-3h) Response After 1 Weeks
Description: as for outcome 8
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to 30 min, 1 h, 2 h, and 3 h relative to dose after 1 week
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | 0.062 (0.024) | 0.264 (0.023) | 0.293 (0.024) | 0.295 (0.023) | 0.321 (0.024)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.202, 95% CI [0.140 to 0.264], Standard Error of Mean 0.032 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.231, 95% CI [0.169 to 0.294], Standard Error of Mean 0.032 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.233, 95% CI [0.172 to 0.295], Standard Error of Mean 0.031 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.259, 95% CI [0.197 to 0.322], Standard Error of Mean 0.032 — Olo 20 mcg qd minus Placebo

16. Secondary Outcome: Peak FEV1 (0-3h) Response After 2 Weeks
Description: as for outcome 8
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose on the first day of randomized treatment (baseline) to 30 min, 1 h, 2 h, and 3 h relative to dose after 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
Liter | 0.079 (0.025) | 0.243 (0.025) | 0.267 (0.025) | 0.282 (0.024) | 0.280 (0.025)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.165, 95% CI [0.101 to 0.228], Standard Error of Mean 0.032 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.189, 95% CI [0.125 to 0.252], Standard Error of Mean 0.032 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.203, 95% CI [0.140 to 0.266], Standard Error of Mean 0.032 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.201, 95% CI [0.137 to 0.265], Standard Error of Mean 0.033 — Olo 20 mcg qd minus Placebo

17. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) (Unsupervised) Area Under Curve 6-12 h (AUC 6-12h) Response at Day 1
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of randomized treatment. Means are adjusted using a model with treatment (trt), baseline as fixed effects and centre as random effect. FEV1 AUC 6-12h was calculated from 6-12 hours post-dose using the trapezoidal rule, divided by the observation time (6h) to report in litres.
Time Frame: baseline and day1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 73 | 75 | 79 | 72 | 73
Liter | 0.019 (0.028) | 0.064 (0.028) | 0.166 (0.027) | 0.195 (0.028) | 0.171 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.2392, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.045, 95% CI [-0.030 to 0.121], Standard Error of Mean 0.039 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.147, 95% CI [0.072 to 0.222], Standard Error of Mean 0.038 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.176, 95% CI [0.099 to 0.253], Standard Error of Mean 0.039 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.152, 95% CI [0.076 to 0.228], Standard Error of Mean 0.039 — Olo 20 mcg qd minus Placebo

18. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) (Unsupervised) Area Under Curve 6-12 h (AUC 6-12h) Response After 1 Week
Description: as for outcome 17
Time Frame: Baseline and 1 week
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 73 | 75 | 79 | 72 | 73
Liter | -0.018 (0.030) | 0.067 (0.030) | 0.156 (0.029) | 0.132 (0.030) | 0.118 (0.030)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0309, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.085, 95% CI [0.008 to 0.162], Standard Error of Mean 0.039 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.174, 95% CI [0.098 to 0.250], Standard Error of Mean 0.039 — Olo 2 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0002, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.150, 95% CI [0.072 to 0.228], Standard Error of Mean 0.040 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0006, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.137, 95% CI [0.059 to 0.214], Standard Error of Mean 0.039 — Olo 20 mcg qd minus Placebo

19. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) (Unsupervised) Area Under Curve 6-12 h (AUC 6-12h) Response After 2 Weeks
Description: as for outcome 17
Time Frame: Baseline and 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 73 | 75 | 79 | 72 | 73
Liter | 0.006 (0.031) | 0.059 (0.031) | 0.135 (0.030) | 0.105 (0.031) | 0.098 (0.031)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.2150, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.053, 95% CI [-0.031 to 0.137], Standard Error of Mean 0.043 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0024, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.129, 95% CI [0.046 to 0.212], Standard Error of Mean 0.042 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0230, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.099, 95% CI [0.014 to 0.184], Standard Error of Mean 0.043 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0333, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.092, 95% CI [0.007 to 0.177], Standard Error of Mean 0.043 — Olo 20 mcg qd minus Placebo

20. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) (Unsupervised) Area Under Curve 6-12 h (AUC 6-12h) Response After 4 Weeks
Description: as for outcome 17
Time Frame: Baseline and 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 73 | 75 | 79 | 72 | 73
Liter | 0.005 (0.031) | 0.058 (0.031) | 0.134 (0.030) | 0.145 (0.032) | 0.094 (0.031)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.2158, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.053, 95% CI [-0.031 to 0.137], Standard Error of Mean 0.043 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0024, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.129, 95% CI [0.046 to 0.212], Standard Error of Mean 0.042 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0013, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.140, 95% CI [0.055 to 0.225], Standard Error of Mean 0.043 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0376, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.090, 95% CI [0.005 to 0.174], Standard Error of Mean 0.043 — Olo 20 mcg qd minus Placebo

21. Secondary Outcome: Weekly Mean Pre-dose Morning Peak Expiratory Flow Rate (PEFR) After 4 Weeks
Description: Baseline PEFR was defined as the mean of the morning PEFR measurements obtained during the week just prior to first dose of randomized treatment.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter/minute
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 78 | 81 | 79 | 86 | 77
Liter/minute | 212.69 (4.431) | 226.39 (4.367) | 233.97 (4.425) | 250.77 (4.244) | 235.75 (4.471)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0211, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 13.705, 95% CI 2-sided [2.070 to 25.340], Standard Error of Mean 5.916 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0004, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 21.285, 95% CI 2-sided [9.581 to 32.990], Standard Error of Mean 5.951 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 38.077, 95% CI 2-sided [26.607 to 49.546], Standard Error of Mean 5.832 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 23.063, 95% CI 2-sided [11.282 to 34.845], Standard Error of Mean 5.990 — Olo 20 mcg qd minus Placebo

22. Secondary Outcome: Weekly Mean Evening PEFR After 4 Weeks
Description: Baseline PEFR was defined as the mean of the evening PEFR measurements obtained during the week just prior to first dose of randomized treatment.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter/minute
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 78 | 81 | 77 | 86 | 75
Liter/minute | 224.65 (4.581) | 235.09 (4.507) | 246.98 (4.621) | 262.88 (4.376) | 250.06 (4.678)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.0973, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 10.446, 95% CI 2-sided [-1.911 to 22.803], Standard Error of Mean 6.283 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0005, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 22.333, 95% CI 2-sided [9.824 to 34.842], Standard Error of Mean 6.360 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 38.232, 95% CI 2-sided [26.054 to 50.409], Standard Error of Mean 6.192 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 25.408, 95% CI 2-sided [12.814 to 38.002], Standard Error of Mean 6.403 — Olo 20 mcg qd minus Placebo

23. Secondary Outcome: Weekly Mean Number of Occasions of Rescue Therapy After 4 Weeks
Description: Weekly mean number of occasions of rescue therapy used per day (PRN salbutamol (albuterol))
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of puffs
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 78 | 81 | 79 | 86 | 77
Number of puffs | 2.914 (0.260) | 2.393 (0.255) | 3.052 (0.258) | 1.949 (0.248) | 2.500 (0.262)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg qd; Test type: Superiority or Other; p = 0.1541, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.520, 95% CI 2-sided [-1.237 to 0.196], Standard Error of Mean 0.364 — Olo 2 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.7065, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.138, 95% CI 2-sided [-0.583 to 0.859], Standard Error of Mean 0.367 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0076, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.964, 95% CI 2-sided [-1.671 to -0.258], Standard Error of Mean 0.359 — Olo 10 mcg qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg qd; Test type: Superiority or Other; p = 0.2626, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.414, 95% CI 2-sided [-1.138 to 0.311], Standard Error of Mean 0.369 — Olo 20 mcg qd minus Placebo

24. Secondary Outcome: Area Under Curve From 0 to 3 Hours (AUC0-3)
Description: AUC0-3 represents the area under the concentration curve of olodaterol and olodaterol glucuronide in plasma from 0 to time t=3.
Time Frame: Baseline and 4 weeks
Population: All evaluable subjects. A subject was considered to be not evaluable if the subject had a protocol violation relevant to the evaluation of pharmacokinetics or had insufficient data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hours/milliliter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 0 | 44 | 58
Picogram*hours/milliliter
  Olodaterol (N=0;0;0;29;58) |  |  |  | 13.3 (37.9) | 20.3 (56.0)
  Olodaterol glucuronide (N=0;0;0;44;44) |  |  |  | 11.6 (52.8) | 21.1 (67.8)

25. Secondary Outcome: Maximum Concentration (Cmax)
Description: Cmax represents the maximum concentration of olodaterol and olodaterol glucuronide in plasma.
Time Frame: Baseline and 4 weeks
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram/milliliter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 54 | 71 | 69
Picogram/milliliter
  Olodaterol (N=0;0;40;71;69) |  |  | 3.58 (51.4) | 5.45 (63.5) | 12.2 (76.0)
  Olodaterol glucuronide (N=0;0;54;71;66) |  |  | 3.94 (97.5) | 5.24 (97.4) | 10.6 (88.1)

26. Secondary Outcome: Time From Dosing to the Maximum Concentration (Tmax)
Description: tmax represents the time from dosing to maximum concentration of olodaterol and olodaterol glucuronide in plasma.
Time Frame: Baseline and 4 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 54 | 71 | 69
hours
  Olodaterol (N=0;0;40;71;69) |  |  | 0.167 [0.0830 to 1.00] | 0.183 [0.0500 to 1.58] | 0.200 [0.0330 to 1.27]
  Olodaterol glucuronide (N=0;0;54;71;66) |  |  | 2.95 [0.0830 to 3.38] | 3.00 [0.0830 to 3.92] | 3.00 [0.0830 to 3.60]

27. Secondary Outcome: Area Under Curve From 0 to 3 Hours at Steady State (AUC0-3,ss)
Description: AUC0-3,ss represents the area under the concentration curve of olodaterol and olodaterol glucuronide in plasma from 0 to time t=3 at steady state.
Time Frame: Baseline and 4 weeks
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hours/milliliter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 55 | 69 | 70
Picogram*hours/milliliter
  Olodaterol (N=0;0;0;63;70) |  |  | NA (NA) — No patients analyzed. | 15.6 (49.9) | 27.7 (64.3)
  Olodaterol glucuronide (N=0;0;55;69;63) |  |  | 9.29 (43.3) | 11.4 (69.0) | 23.9 (68.9)

28. Secondary Outcome: Area Under Curve From 0 to 6 Hours at Steady State (AUC0-6,ss)
Description: AUC0-6,ss represents the area under the concentration curve of olodaterol and olodaterol glucuronide in plasma from 0 to time t=6 at steady state.
Time Frame: Baseline and 4 weeks
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hours/milliliter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 32 | 55 | 69
Picogram*hours/milliliter
  Olodaterol (N=0;0;0;55;69) |  |  | NA (NA) — No patients analyzed. | 29.7 (43.0) | 46.4 (57.3)
  Olodaterol glucuronide (N=0;0;32;50;48) |  |  | 21.4 (40.6) | 25.6 (60.2) | 49.4 (61.0)

29. Secondary Outcome: Area Under Curve From 0 to 24 Hours at Steady State (AUC0-24,ss)
Description: AUC0-24,ss represents the area under the concentration curve of olodaterol and olodaterol glucuronide in plasma from 0 to time t=24 at steady state.
Time Frame: Baseline and 4 weeks
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hours/milliliter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 0 | 39 | 60
Picogram*hours/milliliter
  Olodaterol |  |  |  | 104 (40.9) | 145 (55.1)
  Olodaterol glucuronide |  |  |  | NA (NA) — No patients analyzed. | NA (NA) — No patients analyzed.

30. Secondary Outcome: Maximum Concentration at Steady State (Cmax,ss)
Description: Cmax,ss represents the maximum concentration of olodaterol and olodaterol glucuronide in plasma at steady state.
Time Frame: Baseline and 4 weeks
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram/milliliter
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 60 | 72 | 72
Picogram/milliliter
  Olodaterol (N=0;0;46;72;72) |  |  | 4.02 (46.7) | 7.13 (63.8) | 14.1 (83.4)
  Olodaterol glucuronide (N=0;0;60;72;66) |  |  | 4.90 (49.8) | 5.55 (65.2) | 11.1 (81.0)

31. Secondary Outcome: Time From Dosing to the Maximum Concentration at Steady State (Tmax,ss)
Description: tmax,ss represents the time from dosing to maximum concentration of olodaterol and olodaterol glucuronide in plasma at steady state.
Time Frame: Baseline and 4 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 0 | 0 | 60 | 72 | 72
hours
  Olodaterol (N=0;0;46;72;72) |  |  | 0.192 [0.0830 to 1.02] | 0.200 [0.0500 to 1.02] | 0.200 [0.0830 to 1.00]
  Olodaterol glucuronide (N=0;0;60;72;66) |  |  | 3.00 [0.100 to 6.13] | 3.00 [0.667 to 6.12] | 3.00 [0.000 to 6.03]

32. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, ECG and Physical Examination
Description: Clinical relevant abnormalities for vital signs, ECG and physical examination. Any new or clinically relevant worsening of baseline conditions was reported as adverse events.
Time Frame: 4 weeks
Population: Treated set including all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 79 | 81 | 80 | 86 | 79
participants
  Electrocardiogram QT prolonged | 0 | 1 | 1 | 0 | 2
  Blood creatine phosphokinase increased | 0 | 0 | 0 | 0 | 1
  Gamma-glutamyltransferase increased | 0 | 1 | 0 | 0 | 0
  Atrioventricular block first degree | 0 | 0 | 0 | 0 | 1
  Sinus arrhythmia | 1 | 0 | 0 | 0 | 0
  Tachycardia | 0 | 0 | 1 | 1 | 0
  Palpitations | 0 | 1 | 0 | 0 | 0

33. Secondary Outcome: Laboratory Testing: Average Change From Baseline of Potassium
Description: Laboratory testing: Average change from baseline of potassium measured on test-days. Pre-dose value on test day 1 is the baseline value.
Time Frame: Baseline and day 29
Population: as for baseline characteristics
Measure: Geometric Mean (Inter-Quartile Range); unit: mmol/L
Arm/Group | Placebo | Olo 2 mcg qd | Olo 5 mcg qd | Olo 10 mcg qd | Olo 20 mcg qd
Number analyzed (Participants) | 64 | 73 | 67 | 75 | 66
mmol/L | 0.97 (NA) [0.93 to 1.01] | 0.99 (NA) [0.94 to 1.05] | 0.98 (NA) [0.94 to 1.04] | 0.97 (NA) [0.92 to 1.02] | 0.98 (NA) [0.93 to 1.02]

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Olo 2 mcg: Olodaterol 2 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 5 mcg: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 20 mcg: Olodaterol 20 mcg qd (morning) delivered by the Respimat Inhaler.
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Serious Adverse Events (participants affected / at risk) | 0/79 | 2/81 | 2/80 | 2/86 | 2/79
Other Adverse Events (participants affected / at risk) | 13/79 | 8/81 | 12/80 | 9/86 | 7/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=79) | Olo 2 mcg (N=81) | Olo 5 mcg (N=80) | Olo 10 mcg (N=86) | Olo 20 mcg (N=79)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=79) | Olo 2 mcg (N=81) | Olo 5 mcg (N=80) | Olo 10 mcg (N=86) | Olo 20 mcg (N=79)
Nasopharyngitis (Infections and infestations) | 1 | 2 | 6 | 4 | 2
Headache (Nervous system disorders) | 4 | 3 | 1 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 6 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 2 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.